CLINICAL TRIAL: NCT01125384
Title: Comparison Between Two Methods of Throat Swabbing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: stopped due to protocol mistakes
Sponsor: Meir Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MMC10104-09CTIL
Record Dates: First submitted 2010-05-02; First posted 2010-05-18 (Estimated); Last update posted 2011-08-30 (Estimated); Status verified 2011-08

CONDITIONS: Pharyngitis
MeSH Terms: conditions — Pharyngitis

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- nurse swabbing (No Intervention)
- "accurate" swabbing by a physician (Experimental)
  Interventions: Other: additional swabbing

INTERVENTIONS:
Other: additional swabbing — physician swabs patient's throat according to standard rules before referral of the patient to throat swabbing by nurse.
  Arms: "accurate" swabbing by a physician

SUMMARY:
Throat swabbing is an important instrument in the diagnosis of strep pharyngitis and sometimes the main argument for antibiotic treatment. There is no firm knowledge about an appropriate method of the swabbing for receiving maximal sensitivity. We hypothesize that accurate swabbing from the pus will increase the sensitivity of the swabbing as compared to free swabbing. In order to check this hypothesis we will compare two swabs from the same throat. One that will be taken by a physician specifically from the pass and the second will be taken by a nurse as she used to do it. An increase of 10% of positive results will be accepted as a significant advantage.

ELIGIBILITY:
Inclusion Criteria:

* patients with sore throat, classified 2-3 according to Cantor's criteria

Exclusion Criteria:

* patients on antibiotic treatment
* suspected carriers of streptococcus

Ages: 3 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 500 (Estimated)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
sensitivity of "accurate" swabbing versus sensitivity of habitual nurses' swabbing | 1 year
  Proportion of positive cultures obtained by "accurate" swabbing will be compared to the proportion of positive cultures obtained by nurses' habitual swabbing (as they do it usually).